CLINICAL TRIAL: NCT02526459
Title: The Effect of Birth Plans on Obstetrical Outcomes: a Randomized Control Trial
Brief Title: The Effect of Birth Plans on Obstetrical Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saskatchewan Health Authority - Regina Area (Other)
Responsible Party: Principal Investigator, Rashmi Bhargava, Dr, Saskatchewan Health Authority - Regina Area
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REB-15-31
Record Dates: First submitted 2015-07-31; First posted 2015-08-18 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- birth plan (Experimental): Use of birth plan
  Interventions: Behavioral: Birth plan
- no birth plan (No Intervention): No use of birth plan

INTERVENTIONS:
Behavioral: Birth plan — Patient will receive a birth plan
  Arms: birth plan

SUMMARY:
The study design is a prospective, single institution, randomized control trial in which the introduction of a birth plan is the intervention and a comparison of the rate of Caesarean sections between participants in the control group (no birth plan) and the experimental group (birth plan) is the primary outcome.

DETAILED DESCRIPTION:
The study design is a prospective, single institution, randomized control trial in which the introduction of a birth plan is the intervention and a comparison of the rate of Caesarean sections between participants in the control group (no birth plan) and the experimental group (birth plan) is the primary outcome. In addition, a variety of maternal variables such as epidural use, induction of labour, and excessive blood loss will be collected to be compared between the two groups as it is anticipated that these could have a confounding effect on whether a Caesarean section will be used or not. Furthermore, neonatal outcomes such as birth weight, presence of meconium, and APGAR scores <7 at 5 minutes are also collected for this purpose. A complete list of all collected variable can be found in the data collection form. Patients will be enrolled by Dr. Rashmi Bhargava who sees approximately an average of one patient a day who would be eligible to participate in this project. The investigators aim to enroll a total of about 200 patients from this group over the next 12 to 18 months.

Potential research participants will be approached by the PI, who is a staff obstetrician, during office visits at approximately 34 weeks gestational age. The study will be explained and if the patient is interested in participation, she will receive the study's consent form to take home and look over. It will be stressed to her that she is under no obligation to participate and if she decides not to participate or discontinue participation at a later time, the standard of care she will receive will not be affected. At the following prenatal visit (approximately 36 weeks), patients will bring the completed consent form and concurrently be randomized to either the birth plan group or the control group. Only those randomized to the birth plan group will be provided with a template to assist them in the construction of an individualized birth plan. The staff obstetrician will review and finalize these birth plans and answer any questions the participant may have in the following prenatal visit (approximately 37 weeks). The finalized birth plan will be taken home by the participant, while a copy will be made and faxed from Dr. Bhargava's office to the Labour and Birth Unit at the Regina General Hospital and placed in the participant's file. This way, the birth plan will available for when the participant arrives at RGH for child birth in case she did not bring the original with her. All office visits are scheduled as per normal procedures (standard of care) and are not scheduled solely for the purpose of this research project.

Participants will be randomized in a 1:1 ratio using permuted blocks of 6. A computer generated (SPSS) algorithm will be used to create the randomization sequence table before recruitment starts. Participants will be informed of their allocation at the time of their consent by their obstetrician.

All data will be collected from the participant's chart, except for her rating of childbirth satisfaction, which will be collected through the Mackey Childbirth Satisfaction Rating Scale. This online questionnaire will be completed by patients postpartum using a secure website (FluidSurveys) as an assessment of their satisfaction in labour. To this end, participants are asked to provide their email address on the consent form if they like to complete this questionnaire. Participants will be contacted by email for collection of these surveys about two weeks after child birth. Participants will be required to list their name with their responses so the data can be linked to their other data. As soon as the questionnaire data is collected and the data is linked, the participant's name will be removed and replaced by her study ID.

ELIGIBILITY:
Inclusion Criteria:

* Patient has singleton pregnancy
* Patient has baby with cephalic presentation
* Patient is at less than 34 weeks gestation

Exclusion Criteria:

* Patient has planned Caesarean section
* Patient has planned pre-existing birth plan
* Patient has intrauterine fetal demise
* Patient having a fetus with congenital anomalies
* Existence of intrauterine growth restriction
* Existence of oligohydramnios

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-10; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Caesarean sections (yes/no variable) | 4 weeks
  Was a Caesarean section used to deliver the baby? (yes/no variable abstracted from medical chart)

SECONDARY OUTCOMES:
neonatal outcome: APGAR<7 | 4 weeks
  Scale (abstracted from medical chart)
neonatal outcome: low birth weight | 4 weeks
  Variable abstracted from medical chart
Childbirth Satisfaction (questionnaire) | 4 weeks
  Mackey Childbirth Satisfaction Rating Scale - It rates different satisfaction aspects on a 5-point Likert scale ranging from very dissatisfied to very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Bhargava, MD, Principal Investigator — RQHR
Locations (1):
- Dr Rashmi Bhargava, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No